CLINICAL TRIAL: NCT07026487
Title: Evaluation of The Effect of Music Therapy on Fear of Needle Electromyography
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Hasan Kara, assistant professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HKara4
Record Dates: First submitted 2024-10-16; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Lumbosacral Radiculopathy
Keywords: needle emg; music therapy; electromyography; fear of needle EMG

STUDY DESIGN:
Intervention Model Description: The study will consist of two groups. Intervention group: group receiving treatment with music Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Music therapy will not be given during needle EMG
- Music Group (Experimental): This group will receive music therapy during needle EMG.
  Interventions: Other: Music intervention

INTERVENTIONS:
Other: Music intervention — This group will receive music therapy while performing Needle EMG
  Arms: Music Group

SUMMARY:
Electroneuromyography (ENMG) is a frequently employed methodology in the diagnosis and monitoring of neuromuscular disorders. It encompasses two principal components: nerve conduction studies (NCS) and needle electromyography (EMG). While NST is conducted with the application of electrical stimulation, which may result in mild discomfort, needle EMG is employed for the examination of muscle electrical activity. It is acknowledged that the procedure may cause discomfort, anxiety and fear in patients, which may have an adverse effect on the test results. A variety of methods have been proposed to mitigate discomfort, including oral ibuprofen, cognitive therapy, and topical agents. Music therapy has demonstrated efficacy in alleviating anxiety and pain during numerous medical procedures; however, its impact on pain and anxiety during needle EMG remains unexplored. This study aims to examine the influence of music therapy on pain and anxiety in individuals undergoing needle EMG. To this end, the effects of needle EMG and music therapy on pain and anxiety will be contrasted in two distinct groups.

DETAILED DESCRIPTION:
The objective of this study was to include 58 patients who had been referred to the Erciyes University Faculty of Medicine, Physical Medicine and Rehabilitation, Electroneurophysiology Unit with a prediagnosis of lumbosacral radiculopathy. Following the provision of written informed consent, patients who have agreed to participate in the study will be included. Following the assessment of the inclusion and exclusion criteria, the demographic data of the eligible patients (gender, age, weight, height, body mass index, marital status, occupation, education level) will be recorded on the patient evaluation form.

A comprehensive inquiry will be conducted into the patients' backgrounds, including their medication history, surgical history, preexisting medical conditions, and habits such as smoking and alcohol consumption. Subsequently, the patients will be randomly assigned to either the music treatment group or the control group. In the music group, patients will be provided with the option of listening to a range of relaxing instrumental music, including classical, original, Spanish, jazz, and mystical genres, throughout the EMG procedure. In the control group, no additional procedures will be conducted beyond the routine. To ensure consistency and accuracy, all patients will undergo the same set of measurements before and after the procedure, including the duration of the test, systolic and diastolic blood pressure, and pulse per minute.

The patient's perception of pain during the procedure will be evaluated using the visual analogue scale (VAS), and the State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety Depression Scale (HAD) questionnaires will be completed to assess anxiety levels. Additionally, the level of satisfaction with the procedure, the willingness to undergo the procedure again in the future, the degree of anxiety experienced during the procedure, and the perceived difficulty of the procedure by the physician performing it will be evaluated using a visual analogue scale (VAS) with a range of 0 to 10 points.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years referred to the Electroneuromyography Unit with a prediagnosis of lumbosacral radiculopathy
2. Patients whose cognitive status is sufficient to complete the study and who can be co-operated with

Exclusion Criteria:

1. Individuals with hearing impairment and/or the use of hearing aids
2. Patients with a history of significant neurological or psychiatric illness.
3. Patients with cognitive impairment
4. Patients with a diagnosis of polyneuropathy.
5. Patients receiving pharmacological agents that affect the pain state, including analgesics, antidepressants, and other medications.
6. Individuals who have previously undergone electrodiagnostic studies.
7. Individuals with contraindications for needle EMG, including those with bleeding disorders, anticoagulant use, or active infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | degree of pain during needle EMG, degree of satisfaction with the procedure during needle emg, Whether they are willing to repeat the procedure in the future after needle EMG, anxiety about the procedure: before, during and immediately after procedure
  The patient's perception of pain during the procedure will be assessed with the visual analogue scale (VAS) The degree of satisfaction of the patients with the procedure, their willingness to repeat the procedure in the future, the degree of anxiety during the procedure, and the perceived degree of difficulty in the procedure by the physician performing the procedure will be evaluated with VAS between 0 and 10 points.
State-Trait Anxiety Inventory (STAI) | before and immediately after procedure
Beck Anxiety Inventory | before and immediately after procedure
Hospital Anxiety and Depression Scale | before and immediately after procedure
Systolic-Diastolic Blood pressure | before, during and immediately after procedure
Pulse rate | before, during and immediately after procedure

IPD SHARING:
Plan to Share IPD: No